CLINICAL TRIAL: NCT02400242
Title: A Phase 1a/1b Multicenter, Single-Arm, Open-Label, Dose-Escalation Study to Determine the Maximum Tolerated Dose, Safety, and Preliminary Activity of Oral ACY-241 Alone and in Combination With Pomalidomide and Low-Dose Dexamethasone in Patients With Relapsed or Relapsed-and-Refractory Multiple Myeloma
Brief Title: Study of ACY-241 Alone and in Combination With Pomalidomide and Dexamethasone in Multiple Myeloma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACE-MM-200
Record Dates: First submitted 2015-03-03; First posted 2015-03-27 (Estimated); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — citarinostat; Histone Deacetylase Inhibitors; pomalidomide; Adjuvants, Immunologic; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ACY-241, Pomalidomide, and dexamethasone (Experimental): Open label dosing cohorts will evaluate oral ACY-241 (dosing ranging from 180 mg to 480 mg days 1-21) in combination with oral pomalidomide (4 mg days 1-21), and oral dexamethasone (40 mg qd on days 1, 8, 15, 22).
  Interventions: Drug: ACY-241; Drug: Pomalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: ACY-241 — Dose escalation up to 480 mg administered orally on Days 1-21 of a 28 day cycle.
  Other Names: Histone deacetylase inhibitor
Drug: Pomalidomide — 4 mg qd dosed on days 1-21 of a 28 day cycle
  Other Names: immunomodulatory agent
Drug: Dexamethasone — 40 mg qd on days 1, 8, 15, 22
  Other Names: corticosteriod

SUMMARY:
This is a phase 1a/1b, multicenter, single-arm, open-label, dose escalation study to determine the maximum tolerated dose (MTD) and evaluate the safety and preliminary antitumor activity of ACY-241 for oral administration as monotherapy and in combination therapy with orally administered pomalidomide and low-dose dexamethasone in eligible patients with relapsed or relapsed-and-refractory multiple myeloma (MM).

DETAILED DESCRIPTION:
During phase 1a, patients will receive 1 cycle of ACY-241 monotherapy. Patients who complete the ACY-241 monotherapy cycle without a dose limiting toxicity (DLT) and are clinically stable may continue to phase 1b combination therapy, beginning with Cycle 2. During phase 1b, patients will receive ACY 241 in combination with pomalidomide and low dose dexamethasone at the currently approved pomalidomide dose and schedule. Each cohort of patients in phase 1a and phase 1b will consist of at least 3 patients. The first patient enrolled in each cohort of phase 1a will be observed for 1 week before enrollment of subsequent patients in the cohort. Patients who withdraw consent before entering phase 1b will be replaced. (Replacement patients must complete phase 1a prior to continuing to phase 1b.) Patients who experience a DLT or other unacceptable toxicity in Cycle 1 of phase 1a monotherapy or Cycle 2, the first cycle of phase 1b combination therapy, will be removed from study treatment. An assessment of the safety of treatment will be completed by the Safety Review Committee (SRC) prior to dose-escalation.

ELIGIBILITY:
Key Inclusion Criteria:

* Must have a documented diagnosis of MM and have relapsed or relapsed-and-refractory disease. All patients must have relapsed after having achieved at least stable disease (SD) for at least 1 cycle of treatment to at least 1 prior regimen and then developed progressive disease (PD). Relapsed-and-refractory patients also have documented evidence of PD during or within 60 days of completing last treatment
* Must have undergone prior treatment with at least 2 cycles of lenalidomide and at least 2 cycles of proteasome inhibitor unless not a candidate.
* May have undergone prior treatment with pomalidomide if patient is not refractory to pomalidomide and has previously achieved a response of MR or better to pomalidomide.
* Must have measurable disease (serum M-protein or urine M-protein).
* Must have Eastern Cooperative Oncology Group (ECOG) Performance score of 0, 1, or 2.
* Must be able to take low-dose aspirin, low molecular weight heparin, or other equivalent antithrombotic or anticoagulant daily as prophylactic anticoagulation.

Key Exclusion Criteria:

* Prior therapy with pomalidomide with best response of PD or SD.
* Prior therapy with histone deacetylase (HDAC) inhibitor.
* Any of the following laboratory abnormalities: Absolute neutrophil count(ANC) < 1,000/µL, Platelet count < 75,000/µL or < 50,000/µL for patients in whom ≥ 50% of bone marrow nucleated cells are plasma cells, Hemoglobin < 8 g/dL, Creatinine clearance < 45 mL/min according to Cockcroft-Gault formula. If creatinine clearance calculated from the 24 hour urine sample is ≥ 45 mL/min, patient will qualify for the trial, Aspartate transaminase (AST) or Alanine transaminase (ALT) > 3.0 × Upper Limited Normal (ULN), Serum total bilirubin > 2.0 mg/dL or > 3.0 × ULN for patients with hereditary benign hyperbilirubinaemia.
* Hematologic growth factors are not allowed at screening or during the first cycle of phase 1a or 1b.
* Nonsecretory myeloma or free light chain detected in serum only (ogliosecretory).
* Hypersensitivity to thalidomide, lenalidomide, pomalidomide, or dexamethasone
* Patients who received an allogeneic bone marrow or allogeneic peripheral blood stem cell transplant less than 12 months prior to initiation of study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2015-05-07 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-06-03 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of ACY-241 as monotherapy as assessed by dose limiting toxicities | Cycle 1 (28 days)
Maximum tolerated dose of ACY-241 in combination with pomalidomide and low dose dexamethasone as assessed by dose limiting toxicities | Cycle 2 (28 days)
  First cycle of combination therapy

SECONDARY OUTCOMES:
Frequency and severity of AEs as measured by safety and tolerability | Cycle 1 (28 days)
Single- and multiple-dose peak-plasma concentration | Cycle 1 days 1, 2, 15 and 16
Single- and multiple-dose area under the plasma concentration versus time curve | Cycle 1 days 1, 2, 15 and 16
Change in acetylation of histone and tubulin as a measure of pharmacodynamics | Cycles 1 days 1, 2, 15, 16 and 22
Change in fetal hemoglobin expression as a measure of pharmacodynamics | Cycles 1 days 1, 2, 15, 16 and 22
ACY-241 metabolite concentration in blood samples | Cycles 1 days 1, 2, 15, 16 and 22
Exposure response analyses of potential biomarkers of response. | Cycles 1 days 1, 2, 15, 16 and 22
Frequency and severity of AEs as measured by safety and tolerability in combination | Beginning at Cycle 2 (28 day cycle each) until end of treatment
Change in fetal hemoglobin expression as a measure of pharmacodynamics | Cycle 2 days 1, 2, 15, 16 and 22
Change in acetylation of histone and tubulin as a measure of pharmacodynamics | Cycle 2 days 1, 2, 15, 16 and 22
Single- and multiple-dose area under the plasma concentration versus time curve | Cycle 2 days 1, 2, 15, and 16
Quantification of M-protein as a measure of anti-tumor activity | Day 1 of each cycle beginning at Cycle 2

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (17):
- United States (11):
  - Local Institution - 109, Tucson, Arizona
  - Colorado Blood Cancer Institute, Denver, Colorado
  - University of Miami Medical Center, Miami, Florida
  - Local Institution - 108, Tampa, Florida
  - Local Institution - 103, Atlanta, Georgia
  - Local Institution - 104, Boston, Massachusetts
  - Local Institution - 105, Boston, Massachusetts
  - Local Institution - 101, New York, New York
  - Gabrail Cancer Center Research, Canton, Ohio
  - CTRC at The UT Health Science Center at San Antonio, San Antonio, Texas
  - Local Institution - 111, Seattle, Washington
- France (2):
  - Local Institution - 340, Lille
  - Local Institution - 341, Nantes
- Local Institution - 330, Heidelberg, Germany
- Local Institution - 320, Athens, Greece
- Spain (2):
  - Local Institution - 301, Pamplona
  - Local Institution - 300, Salamanca

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html